CLINICAL TRIAL: NCT03686631
Title: A Behavioral Study of Digital Technology for Improving Post-Operative Incentive Spirometer Adherence
Brief Title: The Digital Incentive Spirometer (DIS): Improving Adherence to Incentive Spirometry
Acronym: DIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Charles Safran, Chief, Division of Clinical Informatics, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018P000230
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Post-Op Infection; Adherence, Patient; Pulmonary Atelectasis; Incentive Spirometry; Post-Op Complication
Keywords: respiratory therapy; Pulmonary Atelectasis; perioperative medicine; incentive spirometry; smartphone
MeSH Terms: conditions — Patient Compliance; Pulmonary Atelectasis; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled randomly into either the passive arm or the smartphone arm prior to their surgery.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The outcomes assessor / statistician will be blinded to which group each patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Arm (No Intervention): This arm uses a passive tracking device to assess the number of times a patient uses their prescribed incentive spirometer.
- Smartphone Arm (Experimental): This arm uses a smartphone connected device and smartphone application to remind and encourage patients to use the spirometer as well as track the number of times they utilize the spirometer.
  Interventions: Behavioral: Smartphone Arm

INTERVENTIONS:
Behavioral: Smartphone Arm — The smartphone arm will have an associated smartphone application, available in kiosk mode, that will remind and encourage patient to utilize the spirometer and provide a "gamified" application for that patient to do so.
  Arms: Smartphone Arm

SUMMARY:
The purpose of the protocol is to assess how incentive spirometer data gathered via a smartphone platform can be utilized to improve participant adherence to prescribed incentive spirometer exercises in the post-operative period. Half of the participants will receive a standard of care incentive spirometer with a passive tracking device while the other half of the participants will receive a smartphone connected device and smartphone with an application that will encourage their use.

DETAILED DESCRIPTION:
This study is a prospective, randomized, participant blinded, single center, clinical trial to ascertain whether a smartphone connected digital incentive spirometer, the Smartpeakflow™, can improve participant adherence to prescribed incentive spirometer exercises. A control group will be given the Beth Israel Deaconess Medical Center (BIDMC) standard Voldyne Incentive Spirometer with an attached microcontroller that will record use of the spirometer. The study group will be given the Smartpeakflow ™ connected to an android motherboard (microcomputer, aka smartphone) running Android OS, that will then record use and store this data on the smartphone itself. Participants will then use an app on the BIDMC provided smartphone to view their usage and receive encouragement to continue using their device. All data on use will be recorded locally and there will be no internet connection or communication with participant through this device at any time.

The study is designed as a technology evaluation to assess feasibility, usability and assess for early impact on our outcome measures. The investigators plan to enroll up to 50 participants to participate in this study.

At the time of enrollment, participants who meet the inclusion criteria, and none of the exclusion criteria, will be asked to opt in to the study. Participants will read information about the study and research staff will explain what it means to "opt in". Prospective participants will be given ample time to read the informed consent form and ask any questions.

Once enrolled, participants will be randomized electronically to either the study group or control group. Participants that are randomized to the control group will have no further training or instructions at the Pre-Anesthesia Testing Clinic. Participants that are in the study group will be instructed on how to use the smartphone application and device which will then be provided to them in the Post Anesthesia Care Unit after their surgery. Both groups will retain and utilize the spirometers throughout their hospital stay, and the devices will be collected by the investigators when the participant is discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Class (ASA) 1-3 patients undergoing elective Surgery at BIDMC requiring Incentive Spirometer use in the post-op period
* Greater than 18 years of age.
* Required to have a Pre-Anesthesia Testing Clinic Appointment
* Able to understand and sign a study consent form
* Able to understand and utilize a smartphone application

Exclusion Criteria:

* Diagnosis of Obstructive Sleep Apnea (OSA), treatment with CPAP or BIPAP for OSA
* Lack of regular smartphone use, or visual, mental or motor impairment that impedes use of smartphone
* Upper extremity surgery resulting in temporary or permanent inability to use two hands with spirometer device
* ASA 4 or greater, any ASA-E status (emergency surgical procedure)
* Suspected or established respiratory infection
* Previous spontaneous pneumothorax
* Severe pulmonary disease, or use of home O2
* Does not speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed post-operative incentive spirometer exercises | Enrollment after patient finishes their surgery and data collection continues until patient is discharged home, or up to 2 weeks, whichever is sooner.
  The primary outcome of the study will be a measure of how adherent the participant has been to the prescribed post-operative incentive spirometer exercises. Participants are prescribed ten breathing exercises per hour using the spirometer and the electronic devices in both arms will record how often the participant utilizes the device, measured on an hourly basis.

SECONDARY OUTCOMES:
Incidence of Post-Operative Pulmonary Complications | Enrollment after patient finishes their surgery and data collection continues until patient is discharged home, or up to 2 weeks, whichever is sooner.
  Pulmonary related complications and events such as radiographic exams, increased utilization of oxygen therapy, use of accessory breathing devices (BiPAP, CPAP). The measure will be dichotomous outcome based on whether event took place or not.
Incidence of post-operative respiratory infection | Enrollment after patient finishes their surgery and data collection continues until patient is discharged home, or up to 2 weeks, whichever is sooner.
  Diagnosis of respiratory infection, such as pneumonia, in the post-operative period. The measure will be dichotomous outcome based on whether event took place or not.
Incidence of clinically relevant complications | Enrollment after patient finishes their surgery and data collection continues until patient is discharged home, or up to 2 weeks, whichever is sooner.
  Diagnosis of clinically relevant complications such as surgical site infection, falls, delerium, or any other non-pulmonary event in the post-operative period. The measure will be dichotomous outcome based on whether event took place or not.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Safran, MD MS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Branson RD. The scientific basis for postoperative respiratory care. Respir Care. 2013 Nov;58(11):1974-84. doi: 10.4187/respcare.02832. PMID 24155356
- [Background] Warner DO. Preventing postoperative pulmonary complications: the role of the anesthesiologist. Anesthesiology. 2000 May;92(5):1467-72. doi: 10.1097/00000542-200005000-00037. No abstract available. PMID 10781293
- [Background] THOREN L. Post-operative pulmonary complications: observations on their prevention by means of physiotherapy. Acta Chir Scand. 1954 May 5;107(2-3):193-205. No abstract available. PMID 13188561
- [Background] Bartlett RH, Gazzaniga AB, Geraghty TR. Respiratory maneuvers to prevent postoperative pulmonary complications. A critical review. JAMA. 1973 May 14;224(7):1017-21. No abstract available. PMID 4574097